CLINICAL TRIAL: NCT01070628
Title: Levodopa Concentration Profile After Repeated Doses of Different Stalevo® Strengths With 3.5 Hours Dosing Frequency; an Open, Randomised, Crossover, Levodopa/Carbidopa Controlled Single Centre Study in Healthy Subjects, Two Parallel Groups
Brief Title: Levodopa Concentration Profile With Stalevo 75/125 mg
Acronym: NEWSTA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Irja Korpela, Clinical Study Manager, Orion Pharma
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2939131
Record Dates: First submitted 2009-11-23; First posted 2010-02-18 (Estimated); Last update posted 2010-08-13 (Estimated); Status verified 2010-08

CONDITIONS: Parkinson's Disease
Keywords: Pharmacokinetic
MeSH Terms: conditions — Parkinson Disease | interventions — Stalevo; Levodopa; Carbidopa; entacapone; carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stalevo (levodopa/carbidopa/entacapone) (Experimental): 125mg or 75mg of levodopa during treatment period 1 in groups 1 and 2 respectively.
  150mg or 100mg of levodopa during treatment period 2 in groups 1 and 2 respectively.
  Interventions: Drug: Stalevo (levodopa/ carbidopa/ entacapone)
- Sinemet (levodopa/carbidopa) (Active Comparator): 150mg or 100mg of levodopa during treatment period 3 in study groups 1 and 2 respectively
  Interventions: Drug: Sinemet (levodopa/carbidopa)

INTERVENTIONS:
Drug: Stalevo (levodopa/ carbidopa/ entacapone) — 150mg, 125 mg, 100mg, 75mg of levodopa q.i.d. in 3.5 h interval
  Other Names: Stalevo
  Arms: Stalevo (levodopa/carbidopa/entacapone)
Drug: Sinemet (levodopa/carbidopa) — 150 or 100 mg levodopa q.i.d. in 3.5 hr interval
  Other Names: Sinemet
  Arms: Sinemet (levodopa/carbidopa)

SUMMARY:
The purpose of this study is to confirm that the dose levels and dosing frequency utilising the new Stalevo strengths would result into more stable levodopa plasma levels. Therefore, it is anticipated that when lower dose of Stalevo is administered after the first higher dose of Stalevo, this would result in equally high levodopa maximum concentration values (Cmax) after each dose throughout the day compared to Cmax after the first dose.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (IC) obtained.
* Good general health ascertained by detailed medical history, and laboratory and physical examinations.
* Finnish speaking males or females, 18-70 years of age inclusive.
* Normal weight defined as body mass index (BMI) 18.5-30.0 kg/m2 (inclusive) (BMI = weight/height2).
* Weight at least 50.0 kg.
* Regular intestinal transit (no recent history of recurrent constipation, diarrhoea, or other intestinal problems).

Exclusion Criteria:

* Evidence of a clinically significant cardiovascular, renal, hepatic, haematological, gastrointestinal, pulmonary, metabolic-endocrine, neurological, urogenital or psychiatric disease as judged by the investigator.
* Any condition requiring regular concomitant treatment (including vitamins and herbal products) or likely to need any concomitant treatment during the study. As an exception, contraceptives or hormone replacement therapy are allowed.
* Intake of any medication that could affect the outcome of the study.
* Any clinically significant abnormal laboratory value or physical finding (including electrocardiogram [ECG]) and vital signs) that may interfere with the interpretation of test results or cause a health risk for the subject if he/she participates in the study, as judged by the investigator.
* Orthostatic hypotension; systolic and diastolic BP and heart rate HR after 3 minutes in supine position and after 3 minutes of standing:
* decrease of ≥ 20 mmHg for systolic BP
* decrease of ≥ 10 mmHg for diastolic BP.
* Strong tendency to motion sickness.
* Known hypersensitivity to the active substance(s) or to any of the excipients of the drug.
* Pregnant or lactating females.
* Females of childbearing potential if they are not using proper contraception (hormonal contraception, intrauterine device (IUD) or surgical sterilization, spermicidal foam/Vagitorie, condom on male partner). Double methods (mentioned above) of contraception is needed during the study. (Note: women of childbearing potential with no current sexual relationship can be included without contraception according to the judgement of the investigator).
* Recent or current (suspected) drug abuse or positive result in the drug abuse test.
* Recent or current alcohol abuse (regular drinking more than 21 units per week for males and more than 16 units per week for females [1 unit = 4 cl spirits or equivalent]).
* Current use of nicotine containing products more than 5 cigarettes (or equivalent)/day and/or inability to refrain from the use of nicotine containing products during the stay at the study centre.
* Use of caffeine containing beverages more than 600 mg of caffeine/day and/or inability to refrain from the use of caffeine containing beverages while at the study centre.
* Blood donation or loss of significant amount of blood within 90 days prior to the first study treatment administration.
* Administration of another investigational treatment within 90 days prior to the first study treatment administration.
* Unsuitable veins for repeated venipuncture or for cannulation.
* Predictable poor compliance or inability to communicate well with the study centre personnel.
* Inability to participate in all treatment periods.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To demonstrate that reduced Stalevo strengths 75 mg and 125 mg following initial 100 mg and 150 mg strengths, will not increase Cmax of levodopa compared to Stalevo or levodopa/carbidopa dosing using equal strengths during the day. | 2-11 weeks

SECONDARY OUTCOMES:
Cmin, AUCo-tau | each subject 3 PK days between 1-6 days

CONTACTS AND LOCATIONS:
Overall Officials: Kimmo Ingman, Principal Investigator — Orion Corporation, Orion Pharma
Locations (1):
- Phase I Unit, Orion Pharma, Espoo, Finland